CLINICAL TRIAL: NCT00297752
Title: A Randomised Multicentre Clinical Trial on the Efficacy of Flammacerium in the Treatment of Facial Burns and the Impact of Facial Burns on Psychosocial Wellbeing
Brief Title: Treatment of Facial Burns With Flammacerium Compared to Flammazine and the Impact of Facial Burns on Psychosocial Wellbeing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Dutch Burns Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO/PO.109
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2009-08

CONDITIONS: Burns
Keywords: facial burns; cerium flammazine; quality of life; randomised clinical trial
MeSH Terms: conditions — Burns | interventions — cerous nitrate, sulfadiazine silver drug combination; Silver Sulfadiazine

ARMS (2):
- 'ceriumnitrate silversulfadiazine (flammacerium) (Active Comparator): facial burns treatment with Cerium nitrate silver sulfadiazine
  Interventions: Drug: ceriumnitrate silversulfadiazine (flammacerium)
- flammazine (Active Comparator): facial burns treatment with silver sulfadiazine
  Interventions: Drug: silversulfadiazine (flammazine)

INTERVENTIONS:
Drug: ceriumnitrate silversulfadiazine (flammacerium) — treatment of patients with facial burns with CE-SSD
  Other Names: CE-SSD
  Arms: 'ceriumnitrate silversulfadiazine (flammacerium)
Drug: silversulfadiazine (flammazine) — treatment of patients with facial burns with SSD
  Other Names: SSD
  Arms: flammazine

SUMMARY:
The face is involved in 40-50% of patients with burns admitted to the Dutch Burn Centres. Scarring of the face as a consequence of burns will often have a detrimental effect on function and aesthetics, and may cause negative effects on psychosocial wellbeing. What the best treatment is for facial burns, minimising scarring, is unclear. Besides that, there is little empirical evidence regarding the impact of facial scarring on psychosocial wellbeing.

In clinical practice good results are felt to be achieved by treatment of facial burns with flammacerium. To substantiate the perceived advantages of flammacerium, its efficacy is compared to flammazine, a current alternative of care. The efficacy of treatment will be assessed in a prospective randomised multicentre clinical trial. Efficacy will be analysed in terms of number of patients requiring surgery and functional and aesthetic outcome.

Apart from medical outcome, this study offers the opportunity to study psychosocial problems associated with facial defects. It is still an unresolved question whether facial scarring causes more or different psychosocial problems. Therefore, self-esteem and quality of life will be examined over time, in relation to depression, posttraumatic stress symptoms and other factors, such as coping style and social support.

By evaluating the efficacy of different treatment strategies, we aim to optimise the standard of care of facial burns. Furthermore, this study wants to shed more light on the psychosocial impact of facial injury. With these results psychosocial professionals will be able to focus on persons at risk and to be better able to meet a patient's personal needs.

ELIGIBILITY:
Inclusion Criteria:

* patients of 18 years of age or older, competent or temporarily incompetent, who are admitted to one of the three dedicated Dutch Burn Centres with burn injuries involving the face

Exclusion Criteria:

* patients not seen within 24 hours postburn
* patients with mental or cognitive deficits that may interfere with providing informed consent
* patients with poor Dutch proficiency
* patients with chemical burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-03; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Regarding the efficacy of treatment | 3 weeks
  time to wound healing
* number of patients requiring surgical excision of their facial burns | 6 weeks
  number of patients requiring surgical treatment for healing of facial burns
Regarding psychosocial impact: | 3 months
  discrepancy between patient and observer scar assessment
* quality of life and self esteem | 6 months post burn
  measurement of self esteem related to scar quality

SECONDARY OUTCOMES:
● quality of scar (patient and observer) | 12 months post burn
  scar assessment by patient and observer scar scale
● scar elasticity, vascularisation and pigmentation, | 12 months post burn
  scar assessment by cutometer and dermaspectrometer
● hypertrophic surface area | 12 months post burn
  scar thickness area
● functional and/or anatomic impairments, | 12 months post burn
  descriptive analysis
● mimic function | 12 months post burn
  physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Nancy van Loey, PhD, Principal Investigator — Association of Dutch Burns Centres; Marianne K Nieuwenhuis, PhD, Principal Investigator — Association of Dutch Burn Centres
Locations (3):
- Netherlands (3):
  - Red Cross Hopsital, Burns Centre, Beverwijk
  - Martini Hospital, Burns centre, Groningen
  - Medical Centre Rijnmond South, Burns centre, Rotterdam

REFERENCES:
- [Derived] Oen IMMH, van Baar ME, Middelkoop E, Nieuwenhuis MK. Effectiveness of cerium nitrate-silver sulfadiazine in the treatment of facial burns: a multicenter, randomized, controlled trial. Plast Reconstr Surg. 2012 Aug;130(2):274e-283e. doi: 10.1097/PRS.0b013e3182589d63. PMID 22842424